CLINICAL TRIAL: NCT02648282
Title: A Phase II Study of GM-CSF Secreting Allogeneic Pancreatic Cancer Vaccine in Combination With PD-1 Blockade Antibody (Pembrolizumab) and Stereotactic Body Radiation Therapy (SBRT) for the Treatment of Patients With Locally Advanced Adenocarcinoma of the Pancreas
Brief Title: Study With CY, Pembrolizumab, GVAX Pancreas Vaccine, and SBRT in Patients With Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J15237; IRB00083132 (Other: JHMIRB)
Record Dates: First submitted 2016-01-05; First posted 2016-01-07 (Estimated); Results first posted 2023-02-28 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Pancreatic Cancer
Keywords: vaccine; immunotherapy; antibody; PD-1; radiation
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cyclophosphamide; pembrolizumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cyclophosphamide, Pembrolizumab, GVAX Pancreas Vaccine, SBRT (Experimental)
  Interventions: Drug: Cyclophosphamide; Drug: GVAX Pancreatic Cancer Vaccine; Drug: Pembrolizumab; Radiation: SBRT

INTERVENTIONS:
Drug: Cyclophosphamide — 200 mg/m2 is to be administered as a 30 minute IV infusion one day prior to GVAX Pancreas Vaccine every 21 days for a total of 8 doses. In the extended treatment phase, eligible patients may receive 200 mg/m2 as a 30 minute IV infusion one day prior to GVAX Pancreas Vaccine every 6 months for an additional 4 doses.
  Other Names: Cytoxan; CY
Drug: GVAX Pancreatic Cancer Vaccine — 2.5E8 cells of each cell line (Panc 6.03/Panc 10.05) for a total of 5E8 cells is to be administered one day after CY and pembrolizumab for a total of 8 doses. In the extended treatment phase, eligible patients may receive 2.5E8 cells of each cell line (Panc 6.03/Panc 10.05) for a total of 5E8 cells administered one day after CY every 6 months for an additional 4 doses.
  Other Names: Pancreas cancer vaccine; Panc 10.05 pcDNA1/GM-Neo, Panc 6.03 pcDNA1/GM-Neo
Drug: Pembrolizumab — 200 mg will be administered as a 30 minute IV infusion one day prior to the GVAX pancreas vaccine every 21 days for a total of 8 doses. In the extended treatment phase, eligible patients may receive 200 mg as a 30 minute IV infusion every 21 days for an additional 9 doses.
  Other Names: MK-3475; KEYTRUDA
Radiation: SBRT — Patients will receive SBRT (6.6 Gy for 5 days) with the second dose of combined immunotherapy (CY/Pembrolizumab/GVAX Pancreas Vaccine).
  Other Names: Stereotactic Body Radiation Therapy

SUMMARY:
This study will be looking at whether combining cyclophosphamide, pembrolizumab (an antibody that blocks negative signals to T cells), GVAX (pancreatic cancer vaccine), and SBRT (focused radiation) is effective (anti-tumor activity) and safe in patients with locally advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced pancreatic adenocarcinoma
2. Patients must have received mFOLFIRINOX or Gemcitabine/ Abraxane based chemotherapy for 4 cycles with last dose of therapy between 2-5 weeks of study enrollment.
3. Age >18 years
4. No metastatic disease
5. ECOG Performance Status of 0 to 1
6. Adequate organ function as defined by study-specified laboratory tests
7. Patients must be able to have fiducials placed for SBRT
8. Must use acceptable form of birth control through the study
9. Signed informed consent form
10. Willing and able to comply with study procedures

Exclusion Criteria:

1. Patients who have been off of mFOLFIRINOX or gemcitabine/abraxane therapy for more than 49 days
2. Patients who have had more than one line of chemotherapy
3. Patients with uncontrolled intercurrent illness, including but not limited to ongoing or active infection, systematic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric condition that would limit compliance with study requirements
4. Patient who have had prior treatment with IL-2, interferon, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-OX-40, anti-CD40, or anti-CTLA-4 antibodies
5. Patients receiving active immunosuppressive agents or chronic use of systemic corticosteroids within 14 days prior to first dose of study drug
6. Patients who have received growth factors, including but not limited to granulocyte-colony stimulating factor (G-CSF), granulocyte macrophage-colony stimulating factor (GM-CSF), erythropoietin, etc. within 14 days of study drug administration
7. Patients with history of any autoimmune disease:inflammatory bowel disease, (including ulcerative colitis and Crohn's Disease), rheumatoid arthritis, systemic progressive sclerosis (scleroderma), systemic lupus erythematous (SLE) autoimmune vasculitis, CNS or motor neuropathy considered to be of autoimmune origin.
8. Patients who have known history of infection with HIV, hepatitis B, or hepatitis C
9. Patients with evidence of interstitial lung disease
10. Patients on home oxygen
11. Patients with oxygen saturation of <92% on room air by pulse oximetry
12. Pregnant or lactating
13. Conditions, including alcohol or drug dependence, or intercurrent illness that would affect the patient's ability to comply with study visits and procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-07-18 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Lee, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- The Sidney Kimmel Comprehensive Cancer at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Cyclophosphamide, Pembrolizumab, GVAX Pancreas Vaccine, SBRT: Cyclophosphamide: 200 mg/m2 is to be administered as a 30 minute IV infusion one day prior to GVAX Pancreas Vaccine every 21 days for a total of 8 doses. In the extended treatment phase, eligible patients may receive 200 mg/m2 as a 30 minute IV infusion one day prior to GVAX Pancreas Vaccine every 6 months for an additional 4 doses.
  GVAX Pancreas Vaccine: 2.5E8 cells of each cell line (Panc 6.03/Panc 10.05) for a total of 5E8 cells is to be administered one day after CY and pembrolizumab for a total of eight doses. In the extended treatment phase, eligible patients may receive 2.5E8 cells of each cell line (Panc 6.03/Panc 10.05) for a total of 5E8 cells administered one day after CY every 6 months for an additional 4 doses.
  Pembrolizumab: 200 mg will be administered as a 30 minute IV infusion one day prior to the GVAX pancreas vaccine every 21 days for a total of 8 doses. In the extended treatment phase, eligible patients may receive 200 mg as a 30 minute IV infusion every 21 days for an additional 9 doses.
  SBRT: Patients will receive SBRT (6.6 Gy for 5 days) with the second dose of combined immunotherapy (CY/Pembrolizumab/GVAX Pancreas Vaccine).
Period: Overall Study
Arm/Group | Cyclophosphamide, Pembrolizumab, GVAX Pancreas Vaccine, SBRT
Started | 58
Completed | 58
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cyclophosphamide, Pembrolizumab, GVAX Pancreas Vaccine, SBRT
Number analyzed (Participants) | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 49
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Distant Metastasis Free Survival (DMFS)
Description: DMFS is defined as the duration of time from start of treatment to identification of distant metastases on imaging or death, whichever occurs first. Estimation based on the Kaplan-Meier curve.
Time Frame: 62 months
Population: All patients who have received at least two doses of immunotherapy and have had their disease re-evaluated with imaging will be considered evaluable for response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cyclophosphamide, Pembrolizumab, GVAX Pancreas Vaccine, SBRT
Number analyzed (Participants) | 54
months | 9.8 [6.3 to 19.4]

2. Secondary Outcome: Number of Participants Experiencing a Grade 3 or Above Treatment Related Toxicities
Description: When calculating the incidence of AEs, each AE (as defined by NCI CTCAE v4.03) will be counted only once for a given subject.
Time Frame: 41 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide, Pembrolizumab, GVAX Pancreas Vaccine, SBRT
Number analyzed (Participants) | 58
Participants | 11

ADVERSE EVENTS:
Time Frame: Serious and Other (Not Including Serious) Adverse Events were evaluated over 41 months. All-cause mortality was evaluated for up to 64 months.
Description: Adverse reporting collection was conducted by regular investigator assessment and laboratory measurements using NCI CTCAE v4.03. During the survival follow-up portion of the trial, participants were evaluated for all-cause mortality past the time frame of treatment and the assessment of adverse events.
Groups:
- Cyclophosphamide, Pembrolizumab, GVAX Pancreas Vaccine, SBRT: Cyclophosphamide: 200 mg/m2 is to be administered as a 30 minute IV infusion one day prior to GVAX Pancreas Vaccine every 21 days for a total of 8 doses. In the extended treatment phase, eligible patients may receive 200 mg/m2 as a 30 minute IV infusion one day prior to GVAX Pancreas Vaccine every 6 months for an additional 4 doses.
  GVAX Pancreas Vaccine: 2.5E8 cells of each cell line (Panc 6.03/Panc 10.05) for a total of 5E8 cells is to be administered one day after CY and pembrolizumab for a total of 8 doses. In the extended treatment phase, eligible patients may receive 2.5E8 cells of each cell line (Panc 6.03/Panc 10.05) for a total of 5E8 cells administered one day after CY every 6 months for an additional 4 doses.
  Pembrolizumab: 200 mg will be administered as a 30 minute IV infusion one day prior to the GVAX pancreas vaccine every 21 days for a total of 8 doses. In the extended treatment phase, eligible patients may receive 200 mg as a 30 minute IV infusion every 21 days for an additional 9 doses.
  SBRT: Patients will receive SBRT (6.6 Gy for 5 days) with the second dose of combined immunotherapy (CY/Pembrolizumab/GVAX Pancreas Vaccine).
Arm/Group | Cyclophosphamide, Pembrolizumab, GVAX Pancreas Vaccine, SBRT
All-Cause Mortality (participants affected / at risk) | 44/58
Serious Adverse Events (participants affected / at risk) | 6/58
Other Adverse Events (participants affected / at risk) | 54/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclophosphamide, Pembrolizumab, GVAX Pancreas Vaccine, SBRT (N=58)
Glucose intolerance (Endocrine disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclophosphamide, Pembrolizumab, GVAX Pancreas Vaccine, SBRT (N=58)
Hypothyroidism (Endocrine disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 8 (9)
Stomach pain (Gastrointestinal disorders) | 5 (7)
Vomiting (Gastrointestinal disorders) | 3 (4)
Chills (General disorders) | 3 (4) — and administrtion site
Fever (General disorders) | 3 (6) — and administration site
Flu like symptoms (General disorders) | 3 (8) — and administration site
Malaise (General disorders) | 4 (4) — and administration site
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (8)
Rash (Skin and subcutaneous tissue disorders) | 8 (11)
Discoloration (Skin and subcutaneous tissue disorders) | 4 (4) — Vaccine Site Reaction
Induration (Skin and subcutaneous tissue disorders) | 54 (173) — Vaccine Site Reaction
Itching (Skin and subcutaneous tissue disorders) | 50 (142) — Vaccine Site Reaction
Redness (Skin and subcutaneous tissue disorders) | 52 (178) — Vaccine Site Reaction
Swelling (Skin and subcutaneous tissue disorders) | 10 (18) — Vaccine Site Reaction
Tenderness (Skin and subcutaneous tissue disorders) | 39 (105) — Vaccine Site Reaction

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT02648282/Prot_SAP_000.pdf